CLINICAL TRIAL: NCT01443559
Title: Phase I Study of Xenogenic Keratoplasty From Porcine Cornea in the Treatment of Infectious Corneal Ulcer
Brief Title: Xenogenic Keratoplasty From Porcine Cornea
Acronym: XKFPC
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: there was not enough patients recruited in this study
Sponsor: Xiamen University (Other)
Responsible Party: Principal Investigator, Zuguo Liu, Dean of Xiamen University Medical School, Xiamen University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EIXM-XKFPC-20110901
Record Dates: First submitted 2011-09-19; First posted 2011-09-29 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Porcine Corneal Xenograph
Keywords: Xenogenic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xenogenic cornea (Experimental)
  Interventions: Genetic: Xenogenic cornea
- human cornea (Active Comparator)
  Interventions: Genetic: homogenic cornea

INTERVENTIONS:
Genetic: Xenogenic cornea — lamellar acellular xenogenic corneas were sterilised by radiation
  Arms: Xenogenic cornea
Genetic: homogenic cornea — homogenic corneas were sterilised by radiation
  Arms: human cornea

SUMMARY:
Acellular porcine cornea is a valid substitution for human cornea because of its similar biological structure, corneal superficial curvature and good histocompatibility toward human. Facing the lack of human cornea donor, it is hypothesised that using acellular lamellar porcine cornea as an alternative of lamellar human cornea to treat infectious corneal ulcer.

DETAILED DESCRIPTION:
Acellular porcine cornea eligibility criteria:

1. fresh porcine cornea,
2. porcine cornea keeping transparent without scar, neovascularization or corneal ulcer,
3. porcine cornea keeping integrative corneal epithelium and endothelium,
4. acellular porcine cornea keeping transparent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe infectious corneal ulcer
* The ulcers can not be controlled with existing antibiotics eye drops or medicine after 1 week treatment
* The infected corneas have risks of penetrating
* The depth of ulcers are less than 400um
* The bridge of the ulcers is away from corneal limbal more than 1mm
* Patients aged 18 or older
* Patients able and willing to sign the informed consent form

Exclusion Criteria:

* Patients with severe infectious corneal ulcer in stable stage
* Patients with corneal ulcers after viruses infection, such as herpes simplex virus
* Patients with corneal ulcers from non-infectious factors, such as toxicity, burn or immunological inflammation
* The ulcers are not cover pupil zone and will not result in visional defect in future
* The depth of ulcer is less than 50um
* Patients has history of keratoplasty surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of rejection in three months after keratoplasty | three months after lamellar keratoplasty
  1. Rate of epithelium rejection Epithelial rejection performances: 1.1 epithelium edema, OR 1.2 epithelium opacity, OR 1.3 epithelial rejection line.
  2. Rate of stroma rejection Stroma rejection performances: 2.1 stroma edema, OR 2.2 stroma opacity, OR 2.3 suture loosing.

SECONDARY OUTCOMES:
Density of regenerative sub-epithelial nerve plex, stromal nerve and stromal keratocytes in vivo confocal microscopy | one year
  Shapes and location:
  1. Sub-epithelial nerve plex is in the depth between 35um to 65um shaping like white thin line with branches in vivo confocal microscopy.
  2. Sromal nerve is in the stromal layer(about 70um to 500um) shaping like white thick trunk with branches in vivo confocal microscopy.
  3. Stromal keratocytes is in the stromal layer like white rod-shape in vivo confocal microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Zuguo Liu, PhD, Study Director — Eye Institute of Xiamen University
Locations (1):
- Xiamen University Affiliated Xiamen Eye Center, Xiamen, Fujian, China